CLINICAL TRIAL: NCT04520165
Title: Effect of Anti-IL5 and Anti-IgE on Alternative Functions of Eosinophils in Severe Asthma
Brief Title: Effect of Biologicals on Alternative Functions of Eosinophils in Severe Asthma
Status: Active, not recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Renaud Louis, Professor, University of Liege
Other Study IDs: 214077
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole induced sputum Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will measure different cytokines in the sputum (interleukin ((IL))-3, granulocyte-macrophage colony-stimulating factor ((GM-CSF)), IL5, IL-13, IL-33, IL-4, IL-25 thymic stromal lymphopoietin ((TSLP)) and eotaxin-1 ) and in the blood to evaluate their ability to predict the response after 6 months and 1 year of treatment with a biologic treatment (anti-IgE, anti-IL5, anti-IL5R) in terms of reduction in exacerbations and corticosteroid use, improvement in Forced expiratory volume in the first second (FEV1) (+200ml), in asthma control (ACQ decrease >0.5, ACT increase >3), in asthma quality of life (increase in AQLQ score > 0.5) and the effect on sputum and blood inflammation.

DETAILED DESCRIPTION:
Severe asthma is observed in 3 to 5% of the asthmatic population and is characterized by a higher rate of exacerbations, poorly controlled asthma and/or a poor lung function. During the last ten years, anti- Immunoglobulin E (IgE) and anti-IL5 (and anti-IL5R) have considerably improved severe asthma status. Treatment with chronic or oral course of corticosteroids is indeed responsible for a lot of side effects. There is however a lack of biomarkers for the prediction of responders to anti-IL5 and anti-IgE.

The investigators have previously found that sputum eosinophil counts are good predictors for improvement in lung function of severe asthmatics using anti-IL5. Sputum cells might not be the only relevant sputum marker for responders to biologics.

The objective is to evaluate the ability of sputum cytokines (protein levels and genes) (IL-3, IL-4, IL-5, IL-13, IL-33 and GM-CSF) to predict the response of severe asthmatics after 6 months and 1 year of treatment with biologics in terms of reduction in exacerbations and corticosteroid use, improvement in FEV1, in asthma control, in asthma quality of life and the effect on sputum and blood inflammation.

Severe asthmatics seen in the Asthma Clinic of CHU of Liege are very well characterized using baseline measure of blood samples, induced sputum, lung function, fractional exhaled nitric oxide (FeNO), asthma control questionnaires (ACT - ACQ) and asthma quality of life questionnaires (AQLQ).

Data on exacerbations during the previous year and current inhaled and oral treatment is also recorded. If FEV1 value is upper than 70% of the predicted value, severe asthmatics also perform a methacholine challenge to evaluate bronchial hyperresponsiveness.

All these measures are repeated after 6 months and 1 year of treatment with anti-IgE and anti-IL5 or anti-IL5R. All the sputum supernatants are stored at -80°C and RNA from sputum cells is also available.

Target sample size: 50 patients

The investigators plan to measure different cytokines in the sputum (IL3, GM-CSF, IL5, IL-13, IL-33, IL-4…) and to evaluate their ability to predict the response after 6 months and 1 year of treatment with different biologics in terms of reduction in exacerbations and corticosteroid use, improvement in FEV1 (+200ml), in asthma control (ACQ decrease >0.5, ACT increase >3), in asthma quality of life (increase in AQLQ score > 0.5) and the effect on sputum and blood inflammation.

Asthmatic patients are recruited through the outpatient clinic and pulmonary rehabilitation centre (CHU, Sart-Tilman, Liege). Asthma is diagnosed as described in the GINA guidelines.

Sputum induction and processing. The sputum is induced and processed as follow: The whole sputum is collected in a plastic container, weighed, and homogenized with three volumes of phosphate-buffered saline (PBS), vortexed for 30 s, and centrifuged at 800g for 10 min at 4° C. The supernatant is separated from the cell pellet by filtration through 2 layers of sterile gauze. A mucolysis is performed by adding an equal volume of 6.5 mM dithiothreitol and the suspension is rocked during 20 min. After a centrifugation of 10 min at 550g, the squamous cells and total cell counts as well as the cell viability are checked by trypan blue exclusion with a manual hemocytometer. The differential leukocyte count is performed on cytospins stained with May-Grünwald-Giemsa on 500 cells.

If the quality criteria (< 30% of squamous cells and viability > 50%) are respected, the cell pellet is mixed with 5 volumes of RNAprotect cell reagent (Qiagen, Hilden, Germany) and kept at -80 °C until RNA extraction.

In total, 50 patient with successful induced sputum supernatant samples before anti-IL-5, anti-IL5R or anti-IgE therapy as well as 6 months and 1 year after will be analyzed. Regarding the sputum cells, patients with good quality samples before and after therapy will allow gene expression analysis.

Immunoassays: The concentrations of the mediators contained in the sputum supernatant are assessed by ELISA Luminex performance assay (R and D systems, Minneapolis, USA) according to the manufacturer's instructions. Spiking experiments of cytokines in sputum supernatants are performed to check that the recovery is between 80% and 120% for all the analytes.

The mediator protein levels will be obtained using Luminex performance XL discovery kit (R and D systems, Minneapolis, USA) for IL-3 and IL-4 (detection limit : 0.09 pg/ml for both). A Luminex high sensitivity performance kit will be used for IL-5, IL-13, IL-33 and GM-CSF. Detection limits are 0.4, 5.1, 1.8 and 1.6 pg/ml respectively.

RNA extraction and RT-qPCR methods Regarding the mediator gene expression levels, primers and probes will all be obtained from IDT (Integrated DNA Technologies, Skokie, IL, USA). PCR efficiencies will be calculated using qbase+ qPCR analysis software (Biogazelle, Zwijnaarde, Belgium). The same program will be used to obtain relative quantitation in gene expression using the 2-∆∆Ct method. HPRT1 and GNB2L1 will be used as reference genes. The patients will be compared with a cohort of 7 healthy subjects.

The Taqman PCR step is performed in 96-well plates and for each sample, 2 µl of cDNA (diluted 1:4) is used in a total reaction volume of 12.5 µl including 500 nM forward primer, 500 nM reverse primer and 250 nM probe for all the tested genes. Every qPCR are realized in duplicate and included non-template controls for each gene. Amplification is performed on the LightCycler 480 Real-Time PCR (Roche, Pleasanton, CA, USA) during 45 cycles as follows: initial activation step: 95 °C for 15 min; denaturation stage: 94 °C for 15 s; annealing and elongation stage: 60 °C for 1 min. All the procedure is done according to the MIQE guidelines for the minimum information required for a qPCR experiment.

Cytokines will also be measured in the blood of a subset of patients.

Study Endpoints

Primary endpoint:

To identify predictors of reduction in exacerbations and in oral corticosteroids dose.

Secondary endpoint:

To identify predictors of improvement in ACQ (-0.5), ACT (+3pts), AQLQ (+ 0.5), sputum eosinophils (<3%), FEV1 (+ 200ml).

Statistical Plan or Data analysis The results will be expressed as mean¡SD or mean¡SEM for continuous variables; median (range) for skewed distributions. For categorical variables, the number of observations and percentages will be given in each category. Comparisons between different subgroups will be performed with a Kruskal-Wallis test or paired t-test / Wilcoxon signed rank test. The Spearman correlation coefficient will be used to measure the association between clinical parameters.

Power calculations indicated a required total sample size of 50 subjects to confirm a change in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Severe asthmatics seen in the Asthma Clinic of CHU of Liege who agree to undergo complete visit at baseline and after 6 months and 1 year of treatment with a biologic and sign informed consent.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe asthmatic patients recruited through the outpatient clinic and pulmonary rehabilitation centre (CHU, Sart-Tilman, Liege). Asthma and severe asthma is diagnosed as described in the GINA guidelines (http://ginasthma.org/).
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2025-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Schleich, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU Liege, Liège, Liege, Belgium

REFERENCES:
- [Background] Moermans C, Deliege E, Pirottin D, Poulet C, Guiot J, Henket M, da Silva J, Louis R. Suitable reference genes determination for real-time PCR using induced sputum samples. Eur Respir J. 2019 Dec 4;54(6):1800644. doi: 10.1183/13993003.00644-2018. Print 2019 Dec. PMID 31601710
- [Background] Delvaux M, Henket M, Lau L, Kange P, Bartsch P, Djukanovic R, Louis R. Nebulised salbutamol administered during sputum induction improves bronchoprotection in patients with asthma. Thorax. 2004 Feb;59(2):111-5. doi: 10.1136/thorax.2003.011130. PMID 14760148
- [Background] Schleich F, Graff S, Nekoee H, Moermans C, Henket M, Sanchez C, Paulus V, Guissard F, Donneau AF, Louis R. Real-word experience with mepolizumab: Does it deliver what it has promised? Clin Exp Allergy. 2020 Jun;50(6):687-695. doi: 10.1111/cea.13601. Epub 2020 Apr 14. PMID 32198794
- [Background] Moermans C, Brion C, Bock G, Graff S, Gerday S, Nekoee H, Poulet C, Bricmont N, Henket M, Paulus V, Guissard F, Louis R, Schleich F. Sputum Type 2 Markers Could Predict Remission in Severe Asthma Treated With Anti-IL-5. Chest. 2023 Jun;163(6):1368-1379. doi: 10.1016/j.chest.2023.01.037. Epub 2023 Feb 3. PMID 36740095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was performed at the CHU of Liege, Belgium, between 2014 and 2021
Pre-assignment Details: Inclusion criteria included a diagnosis of asthma defined by the Global Initiative for Asthma (http://ginasthma.org/), severe asthma was defined according to European Respiratory Society (ERS)/ American Thoracic Society (ATS) criteria 1. The treatment was stable for all patients at the time of the sampling and the time between baseline and the next evaluation was in average one year
Groups:
- Remission /Not: Fifty-two severe asthmatics initiated with an anti-IL-5 (51 with Mepolizumab and one with Reslizumab) were recruited from our asthma clinic. Remission was defined as patients combining after the instauration of the biotherapy: no oral corticosteroids, no exacerbation, ACQ lower than 1.5 and/or asthma control test (ACT) greater than 19 and, a FEV1 greater than 80% predicted and/or an improvement of FEV1 at least 10% from baseline and a blood eosinophil count lower than 300 cells/microliter.
Period: Overall Study
Arm/Group | Remission /Not
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remission /Not
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — remission group
  years | 48 (18)
Sex: Female, Male [Count of Participants; unit: Participants] — female/male
  Participants
    Female | 29
    Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 52
Region of Enrollment [Number; unit: participants] — CHU Liege Belgium
  participants
    Belgium | 52

OUTCOME MEASURES:

1. Primary Outcome: Presence of Prognostic Markers of Remission in the Sputum Cell Compartment or Not
Description: Remission was defined as patients combining after the instauration of the biotherapy: no oral corticosteroids, no exacerbation, ACQ lower than 1.5 and/or asthma control test (ACT) greater than 19 and, a FEV1 greater or equal to 80% predicted and/or an improvement of FEV1 greater or equal to 10% and a blood eosinophil count lower than 300 cells/microliter.
  Markers of remission in the sputum cell profile were investigated.
Time Frame: 1 year follow-up
Population: To compare groups, baseline characteristics were compared with Mann-Whitney U test
Measure: Median (Inter-Quartile Range); unit: cells/g
Groups:
- Remission: Remission was defined as patients combining after the instauration of the biotherapy: no oral corticosteroids, no exacerbation, ACQ lower than 1.5 and/or asthma control test (ACT) greater than 19 and, a FEV1 greater than 80% predicted and/or an improvement of FEV1 at least 10% from baseline and a blood eosinophil count lower than 300 cells/microliter.
- No Remission: patients that did not fulfilled the remission criteria
Arm/Group | Remission | No Remission
Number analyzed (Participants) | 11 | 41
cells/g
  Sputum eosinophil count | 494000 [235000 to 1663000] | 156000 [16000 to 362000]
  Sputum neutrophil count | 798000 [437000 to 3689000] | 943000 [544000 to 2604000]
  Sputum macrophage count | 526000 [296000 to 988000] | 193000 [92000 to 504000]
  Sputum lymphocyte count | 32000 [7000 to 144000] | 4000 [0 to 31000]
Statistical Analysis 1: Comparison: Remission vs No Remission; The baseline parameters in each group were compared with Mann-Whitney U test was performed; Test type: Equivalence — if p<0.05 than the null hypothesis was considered as wrong and groups differed for the analysed parameter; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Presence of Prognostic Markers (Mediators) of Remission in the Sputum or Not
Description: Remission was defined as patients combining after the instauration of the biotherapy: no oral corticosteroids, no exacerbation, ACQ lower than 1.5 and/or asthma control test (ACT) greater than 19 and, a FEV1 greater or equal to 80% predicted and/or an improvement of FEV1 greater or equal to 10% and a blood eosinophil count lower than 300 cells/microliter.
  Markers ( inflammatory mediators) of remission in the sputum were investigated.
Time Frame: 1 year follow-up
Population: To compare groups, baseline characteristics were compared with Mann-Whitney U test
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Remission | No Remission
Number analyzed (Participants) | 11 | 41
pg/ml
  Eotaxin-1 | 71 [56 to 204] | 54 [0 to 87]
  TSLP | 3.2 [2.4 to 6.5] | 2.2 [1.0 to 3.6]
  IL-5 | 11.5 [3.5 to 22.2] | 2.7 [1.3 to 4.8]
  EPX | 183000 [129000 to 342000] | 48000 [30000 to 99000]
  IgE | 1200 [400 to 2400] | 400 [300 to 600]

3. Secondary Outcome: is EPX in the Sputum of Prognostic Marker of ACT Improvement in the Sputum or Not ?
Description: ACT improvement = greater than 19 post-treatment, EPX = Eosinophil peroxidase in the sputum supernatant
Time Frame: 1 year follow-up
Population: To compare groups, baseline characteristics were compared with Mann-Whitey U test
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Remission | No Remission
Number analyzed (Participants) | 11 | 41
ng/ml | 129 [47 to 241] | 48 [30 to 148]
Statistical Analysis 1: Comparison: Remission vs No Remission; The baseline parameters in each group were compared with Mann-Whitney U test was performed; Test type: Equivalence — if p<0.05 than the null hypothesis was considered as wrong and groups differed for the analysed parameter; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Is IL-5 in the Sputum a Prognosis Marker for Improvement of FEV1 Post-treatment or Not ?
Description: improvement of FEV1 = at least 10% post-treatment IL-5 = interleukin 5 measured in the sputum supernatant
Time Frame: 1 year follow-up
Population: To compare groups, baseline characteristics were compared with Mann-Whitney U test
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- No Remission: patients who did not fulfilled the remission criteria after one year of treatment
Arm/Group | Remission | No Remission
Number analyzed (Participants) | 11 | 41
pg/ml | 9 [2 to 22] | 3 [1 to 5]
Statistical Analysis 1: Comparison: Remission vs No Remission; The baseline parameters in each group were compared with Mann-Whitney U test was performed; Test type: Equivalence — if p<0.05 than the null hypothesis was considered as wrong and groups differed for the analysed parameter; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: In this study, we assessed the prognosis factors of remission after anti IL-5 therapy, the goal was not to assess the impact of the therapy itself on the patient condition.
Arm/Group | Remission /Not
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04520165/Prot_SAP_000.pdf